CLINICAL TRIAL: NCT02800317
Title: Primary Radioactive Iodine Seed Localisation in the Axilla in Axillary Node Positive Breast Cancer Combined With Sentinel Node Procedure (RISAS) Following Neoadjuvant Chemotherapy
Brief Title: RISAS Procedure in Node Positive Breast Cancer Following NAC
Acronym: RISAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Collaborators: Amphia Hospital (Other); Maastricht University Medical Center (Other); UMC Utrecht (Other)
Responsible Party: Principal Investigator, L.B. Koppert, MD, PhD, Erasmus Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2015-8023; NCT02792101 (obsolete NCT alias)
Record Dates: First submitted 2016-06-07; First posted 2016-06-15 (Estimated); Last update posted 2022-02-10 (Actual); Status verified 2022-02

CONDITIONS: Breast Neoplasm; Neoadjuvant Therapy; Axillary Lymph Nodes; Pathological Complete Response
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RISAS (Experimental): All patients will undergo RISAS procedure, followed by axillary lymph node dissection in a one-step surgical procedure.
  Interventions: Procedure: RISAS

INTERVENTIONS:
Procedure: RISAS — RISAS procedure contains Radioactive Iodine Seed localisation in the Axilla in axillary node positive breast cancer combined with a Sentinel node procedure.

SUMMARY:
Chemotherapy in clinically node positive breast cancer patients is increasingly administrated in a neoadjuvant setting. The standard treatment regimen in these cases is then: neoadjuvant chemotherapy (NAC) followed by breast surgery and an axillary lymph node dissection (ALND). NAC results in axillary pathologic complete response (pCR) in 1 out of 3 patients, indicating a complete absence of axillary metastases after completion of NAC. In such events, ALND can be regarded as overtreatment that creates unnecessary morbidity. Less invasive axillary surgery which can accurately assess axillary pCR is therefore preferred over standard ALND in all patients. In case of detection of remaining axillary lymph node metastases by this less invasive axillary surgical procedure, completion axillary treatment is standard of care.

The novel RISAS procedure is introduced as a possible less invasive axillary staging procedure. RISAS procedure contains Radioactive Iodine Seed localisation in the Axilla in axillary node positive breast cancer combined with a Sentinel node procedure. The iodine seed in the axillary lymph node metastasis will be placed prior to start of NAC.

ELIGIBILITY:
Inclusion Criteria:

* Female patient with pathologically confirmed axillary lymph node positive invasive primary breast cancer, treated with neoadjuvant chemotherapy
* Willing and able to undergo all study procedures.
* Has personally provided written informed consent.

Exclusion Criteria:

* Age < 18
* Pregnancy or lactation
* Contra indications for undergoing iodine seed placement or sentinel lymph node biopsy, such as allergic reaction on iodine, 99m Technetium or patent blue.
* Recurrent breast cancer
* Previous axillary surgery or radiotherapy
* Patients with periclavicular lymph node metastases (cN3)
* Patients with advanced breast cancer (i.e. patients with distant metastases, treated without any furter surgical procedures)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Actual)
Dates: Start 2017-03-30 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2021-12-03 (Actual)

PRIMARY OUTCOMES:
Identification rate and accuracy (sensitivity, negative predictive value (NPV) and false negative rate (FNR)) of RISAS-procedure for identifying axillary pCR, with 95% confidence intervals will be calculated. | Participants will be followed from the moment of first out-hospital clinic visit untill final breast surgery, an expected average of 4 months.

SECONDARY OUTCOMES:
The identification rate and accuracy (sensitivity, NPV and FNR) of both techniques used in RISAS-procedure (i.e. SLNB and MARI) for identifying axillary pCR, will be calculated separately as well. | Participants will be followed from the moment of first out-hospital clinic visit untill final breast surgery, an expected average of 4 months.

CONTACTS AND LOCATIONS:
Overall Officials: Linetta B Koppert, MD, PhD, Principal Investigator — Erasmus Medical Center; Ernest JT Luiten, MD, PhD, Principal Investigator — Amphia Hospital; Marjolein L Smidt, MD, PhD, Principal Investigator — Maastricht University Medical Center
Locations (14):
- Netherlands (14):
  - Wilhelmina Hospital, Assen
  - Amphia Hospital, Breda
  - Albert Schweitzer Hospital, Dordrecht
  - Martini Hospital, Groningen
  - Zuyderland Medical Center, Heerlen
  - Hospital Group Twente, Hengelo
  - Treant, Hoogeveen
  - Maastricht University Medical Center, Maastricht
  - Bravis Hospital, Roosendaal
  - Erasmus Medical Center, Rotterdam
  - Ikazia Hospital, Rotterdam
  - Maasstad Hospital, Rotterdam
  - Franciscus Gasthuis & Vlietland, Schiedam
  - University Medical Center Utrecht, Utrecht

REFERENCES:
- [Background] van Nijnatten TJA, Simons JM, Smidt ML, van der Pol CC, van Diest PJ, Jager A, van Klaveren D, Kam BLR, Lobbes MBI, de Boer M, Verhoef K, Koppert LB, Luiten EJT. A Novel Less-invasive Approach for Axillary Staging After Neoadjuvant Chemotherapy in Patients With Axillary Node-positive Breast Cancer by Combining Radioactive Iodine Seed Localization in the Axilla With the Sentinel Node Procedure (RISAS): A Dutch Prospective Multicenter Validation Study. Clin Breast Cancer. 2017 Aug;17(5):399-402. doi: 10.1016/j.clbc.2017.04.006. Epub 2017 Apr 19. PMID 28487053
- [Derived] van Amstel FJG, de Mooij CM, Simons JM, Mitea C, van Diest PJ, Nelemans PJ, van der Pol CC, Luiten EJT, Koppert LB, Smidt ML, van Nijnatten TJA; REFINE Study Group. Disease extent according to baseline [18F]fluorodeoxyglucose PET/CT and molecular subtype: prediction of axillary treatment response after neoadjuvant systemic therapy for breast cancer. Br J Surg. 2024 Aug 30;111(9):znae203. doi: 10.1093/bjs/znae203. PMID 39302345